CLINICAL TRIAL: NCT01341613
Title: Efficacy of a Supplement Capsule Containing L. Reuteri Cardioviva™ on Managing Cholesterol Levels in Hypercholesterolemic Humans
Brief Title: Efficacy of Cardioviva™ Probiotic Supplement Capsule Formulation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Micropharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP-0110
Record Dates: First submitted 2011-04-22; First posted 2011-04-26 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-11

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cardioviva™ supplement capsule (Experimental)
  Interventions: Dietary Supplement: Cardioviva™ supplement capsule
- Placebo capsule (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo capsule

INTERVENTIONS:
Dietary Supplement: Cardioviva™ supplement capsule — Twice per day (BID), 9 weeks
  Arms: Cardioviva™ supplement capsule
Dietary Supplement: Placebo capsule — Twice per day (BID), 9 weeks
  Arms: Placebo capsule

SUMMARY:
Background: It is becoming increasingly clear that individuals from all corners of the globe use probiotic dietary approaches to enhance health. More recently, probiotics have shown promise in treating a variety of disease states, due to improved strain selection, stability and delivery technologies.

Objective: The purpose of this study is to determine the lipid lowering efficacy of a probiotic supplement capsule containing Lactobacillus reuteri Cardioviva™, taken twice per day over 9 weeks, in subjects with hypercholesterolemia.

Design: The study design is a double-blinded, placebo-controlled, randomized, parallel-arm, multi-centre study. The study will last a total of 13 weeks, including a 2-week wash-out period, a 2-week run-in period and a 9 week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, aged 20 to 75 years (bounds included)
* LDL-Cholesterol above 3.4 mmol/L (<15% variation between visits V1 and V2-1)
* TG levels below 4.0 mmol/L (checked at visits V0 and V2-1)
* BMI range will be 22 to 32 kg/m²
* Subject understands and accepts to follow the dietary recommendations advisable for hypercholesterolemic patients (according to NCEP-ATP III guidelines)
* For subjects on statin monotherapy: dosage of statin must be stable for at least 3 months prior to the study beginning (15-20% of all subjects)
* Judged by the investigators as compliant (>80%) with product consumption (check at V2-1), and motivated
* Signed informed consent form prior to inclusion in the study
* Note: Subjects will be permitted to take stable doses of thyroid hormone and anti-hypertensive agents, as long as these are continued equivalently throughout the duration of study
* For female subjects: effective contraceptive methods used

Exclusion Criteria:

* Use of cholesterol lowering prescription drugs other than statin monotherapy within the last 6 months
* Use of plant sterols, omega 3, fish oil, soy protein, soluble oat fiber, psyllium seed husk, or other cholesterol lowering non-prescription food supplements within last 3 months
* History of chronic use of alcohol (>2 drinks/d)
* Use of systemic antibodies, corticosteroids, androgens, or phenytoin
* Subject having experienced any cardiovascular event (Myocardial infarction, coronary artery bypass, or other major surgical procedures) in the last 6 months
* Diabetic subject (Type I or Type II)
* Subject receiving systemic treatment or topical treatment likely to interfere with evaluation of the study parameters
* Subject currently involved in a clinical trial or in an exclusion period following participation in another clinical trial
* History of angina, congestive heart failure, inflammatory bowel disease, pancreatitis, gastrointestinal, renal, pulmonary, hepatic or biliary disease, or cancer (evidence of active lesions, chemotherapy or surgery in the past year)
* Chronic user of probiotics or fibre laxative (greater than 2 doses/wk), or stimulant laxatives
* History of eating disorders
* Exercise greater than 15 miles/wk or 4,000 kcal/wk
* For female subjects: Pregnancy, breast feeding, or intent to get pregnant

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2011-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the percent difference in LDL-cholesterol from baseline to endpoint comparing subjects receiving treatment and placebo | 9 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- APharma s.r.o., Prague, Czechia

REFERENCES:
- [Derived] Jones ML, Martoni CJ, Ganopolsky JG, Sulemankhil I, Ghali P, Prakash S. Improvement of gastrointestinal health status in subjects consuming Lactobacillus reuteri NCIMB 30242 capsules: a post-hoc analysis of a randomized controlled trial. Expert Opin Biol Ther. 2013 Dec;13(12):1643-51. doi: 10.1517/14712598.2013.833601. Epub 2013 Sep 28. PMID 24074303
- [Derived] Jones ML, Martoni CJ, Prakash S. Letter to the editor regarding the report of Duboc et al: Connecting dysbiosis, bile-acid dysmetabolism and gut inflammation in inflammatory bowel disease. Gut. 2013 Apr;62(4):654-5. doi: 10.1136/gutjnl-2012-303867. Epub 2012 Nov 12. No abstract available. PMID 23148122
- [Derived] Jones ML, Martoni CJ, Di Pietro E, Simon RR, Prakash S. Evaluation of clinical safety and tolerance of a Lactobacillus reuteri NCIMB 30242 supplement capsule: a randomized control trial. Regul Toxicol Pharmacol. 2012 Jul;63(2):313-20. doi: 10.1016/j.yrtph.2012.04.003. Epub 2012 Apr 25. PMID 22561556